CLINICAL TRIAL: NCT00945178
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Two-part Study to Assess Safety, Tolerability, Pharmacokinetics of Orally Administered AZD1386
Brief Title: Double-blind Placebo-controlled 2-part Study Assessing the Safety, Tolerability and PK of AZD1386 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to results in another study (NCT00878501).
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D5090C00021; EudraCT No.: 2009-012114-43
Record Dates: First submitted 2009-07-17; First posted 2009-07-24 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Healthy; Pharmacokinetics
MeSH Terms: interventions — AZD1386; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A: A (Experimental): AZD1386
  Interventions: Drug: AZD1386
- Part A: B (Experimental): Placebo for AZD1386
  Interventions: Drug: Placebo for AZD1386
- Part B: A (Experimental): Naproxen
  Interventions: Drug: Naproxen
- Part B: B (Experimental): Placebo for Naproxen
  Interventions: Drug: Placebo for Naproxen

INTERVENTIONS:
Drug: AZD1386 — Single ascending and multiple (twice daily) oral doses, capsule
  Arms: Part A: A
Drug: Placebo for AZD1386 — Single ascending and multiple (twice daily) oral doses, capsule
  Arms: Part A: B
Drug: Naproxen — Tablet, single oral dose, 500mg
  Arms: Part B: A
Drug: Placebo for Naproxen — Tablet, single oral dose
  Arms: Part B: B

SUMMARY:
The study will investigate how a new formulation of the study drug is absorbed, metabolised and distributed through the body, as well as its safety and tolerability in higher doses when given as single and multiple doses and as a single dose in the presence and absence of naproxen.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Healthy male and female (of non childbearing potential)
* Body Mass Index (BMI) of ≥19 to ≤28 kg/m2 and a weight of ≥50 to ≤100 kg

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder in the opinion of the investigator.
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, ECG, safety lab) | Assessments performed at frequent timepoints (predose then ranging from 15 minutes to every 12 hours) on Days -1 to Day 3 (Part A: treatment period 1 and Part B) or Day-1 to Day 9 (Part A: treatment period 2) and at follow-up 4-14 days after discharge.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD1386 in plasma | Assessments performed at frequent timepoints (predose then ranging from 15 minutes to every 12 hours) on Days -1 to Day 3 (Part A: treatment period 1 and Part B) or Day-1 to Day 9 (Part A: treatment period 2).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leff, Study Director — AstraZeneca Pharmaceuticals, Wilmington, UK; Dr. Tania Hugo, Principal Investigator — PAREXEL Early Phase Clinical Unit, London UK.
Locations (1):
- Research Site, Harrow, United Kingdom